CLINICAL TRIAL: NCT07135635
Title: The Value of Doppler Indices Of Middle Cerebral Artery For Prediction Of Fetal Outcome In Pregnant Women With Anemia
Brief Title: Middle Cerebral Artery Doppler( MCA-PSV) & Perinatal Outcome
Status: Enrolling by invitation | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Mahmoud, specialist at elhelal hospital for health insurance, Sohag University
Other Study IDs: Soh-Med-25-5-1 MD
Record Dates: First submitted 2025-08-05; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Anemia During Pregnancy; Anemia Complicating Pregnancy; Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

INTERVENTIONS:
Diagnostic Test: Middle Cerebral Artery doppler — All cases of pregnant women diagnosed with anemia at 3rd trimester will have baseline assessment of history, clinical examination, HB level, obstetric ultrasonography done then they will have Middle Cerebral Artery Doppler done to assess correlation between MCA Doppler indices & neonatal outcomes. Then appropriate treatment of anemia will be taken.

SUMMARY:
can we predict neonatal outcome by the results of 3rd trimester MCA Doppler Indices In pregnant women with anemia?? --- the aim of this study is to evaluate values of MCA Doppler indices in determining fetal outcome in pregnant women with anemia.

DETAILED DESCRIPTION:
This Cross_ sectional study will be performed At OBS/ GYN Department Sohag University Hospital for 1 year duration between February 2025 to February 2026.

All cases of pregnant women diagnosed with anemia at 3rd trimester will have baseline assessment of history, clinical examination, HB level, obstetric ultrasonography done then they will have Middle Cerebral Artery Doppler done to assess correlation between MCA Doppler indices & neonatal outcomes. Then appropriate treatment of anemia will be taken.

Doppler indices and placental weight.

ELIGIBILITY:
Inclusion Criteria:

- (1) Pregnant women diagnosed with anemia at 3rd trimester with hemoglobin level ≤ 11 g/dl.

(2) Singleton pregnancy.

Exclusion Criteria:

1. Multifetal pregnancy.
2. Fetal Anomalies.
3. Any other maternal systemic diseases other than anemia as DM, Preeclampsia, Autoimmune disease.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women with anemia in sohag university hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Third Trimester Middle Cerebral artery Doppler ( MCA -PSV). | 1 year
Assess correlation between MCA Doppler indices and neonatal Hemoglobin level | 1 year

SECONDARY OUTCOMES:
Assess correlation between MCA Doppler indices and neonatal weight. | 1 year
Assess correlation between MCA Doppler indices and NICU admission. | 1 year
Assess correlation between MCA Doppler indices and APGAR Score. | 1year
Assess correlation between MCA Doppler indices and placental weight. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Ahmed professor of obstetrics & gynecology sohag university, professor, Principal Investigator — sohag faculty of medecine
Locations (1):
- Faculty of Medicine- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes